CLINICAL TRIAL: NCT05034913
Title: Use of Digital Photography to Estimate Anthropometric Measurements in Children
Brief Title: Digital Photography to Estimate Anthropometric Measurements in Children
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Initial data analysis prior to full enrollment showed that concept was not valid.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Siobhan T. Pittock, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-011901
Record Dates: First submitted 2021-08-31; First posted 2021-09-05 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Photography to Measure Children's Height, Wrist Circumference, and Abdominal Circumference (Experimental): Subjects will be given instructions on how to take two photographs at home and submit them securely. Subjects will also be given instructions on how to measure height, wrist circumference, and waist circumference and submit this data to the research team.
  Interventions: Other: Digital photography measurements

INTERVENTIONS:
Other: Digital photography measurements — The participant will be instructed to take off any thick outer layers and leave on shirt and pants. Tops will be gathered to make cloth tight to body. The participant will stand next to an 8 ½" x 11" piece of paper taped to a wall, to use as a reference for linear regression calculations.

SUMMARY:
The purpose of this study is to see if photos taken from home can accurately let physicians know the height, abdominal circumference, and wrist circumference of children, and how these measurements relate to in-person measurements.

DETAILED DESCRIPTION:
This study will occur in two distinct parts. Children age 2-18 who present to Mayo for an outpatient clinic appointment will be considered for participation in the study. Patients eligible for the study will receive a portal message the day prior to their appointment informing them of the option to take place in the study as well as instructions on how to measure height, abdominal circumference, and wrist circumference, and how to obtain and submit digital photographs. Participants can submit photographs and home measurements either before or after the in clinic measurements and photographs have been obtained. Those willing to participate will sign a parental consent form and a child assent form. Consent and assent forms can be seen in the supplemental documents.

At Home Participants will be given written instructions asking for 2 photographs to be submitted via the patient portal and for measurements of height, abdominal circumference, and wrist circumference to be obtained using a home tape measure. Detailed patient instructions will be shared.

Study Visit

Traditional Anthropometric Measurements Participant will have a height measurement using a calibrated stadiometer, a weight measurement taken on a scale, a waist circumference taken at the umbilicus, and a wrist circumference will be taken while seated on the dominant wrist over the Lister tubercle of the radius and over the distal ulna. Participants 5 years of age and older who are 90cm and greater will have body composition assessed by impedance. Bioelectrical impedance is not in any way uncomfortable and does not expose the participant to any radiation. Participant measurements will be recorded in the patient record and a secure excel document or in RedCap. Recruited patient's medical record number (MRN) will be documented in a secure excel document or in RedCap.

Digital Photography Measurements The participant will be instructed to take off any thick outer layers and leave on shirt and pants. Tops will be gathered to make cloth tight to body. The participant will stand next to an 8 ½" x 11" piece of paper taped to a wall, to use as a reference for linear regression calculations. The participant will have a photograph taken in the "Frankfurt plane" with lower border of the eyes in line with the external ear canal, palms facing forward and arms to the side, while taking a deep breath at the time of the photograph to have optimal stretching. A photograph will be taken from the side in the sagittal plane with palms facing down and arms outstretched in front of the patient while taking a deep breath at the time of the photograph for optimal stretching. These photos will be taken by a trained member of the research team.

ELIGIBILITY:
Inclusion Criteria:

* Children age 2-18 years old.
* Seen on Mayo 16 for an outpatient clinic appointment.

Exclusion Criteria:

* Participant unable to stand for stadiometer height
* Pregnant patients

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
Height | 1 day
  Measured in cm
Abdominal circumference | 1 day
  Measured in cm
Wrist circumference | 1 day
  Measured in cm

CONTACTS AND LOCATIONS:
Overall Officials: Siobhan Pittock, M.B., B.Ch,, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials